CLINICAL TRIAL: NCT07103382
Title: Efficacy and Safety of Attapulgite in Patients With Obesity: An Exploratory Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yang Xiao, Associate Professor, Department of Metabolism and Endocrinology, Institute of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital, Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025 Attapulgite
Record Dates: First submitted 2025-07-10; First posted 2025-08-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: attapulgite; obesity; placebo-controlled study; randomized controlled trial
MeSH Terms: conditions — Obesity | interventions — attapulgite

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attapulgite (Experimental): Attapulgite capsules (0.4-0.5 g) were administered at a dose of 3 capsules twice daily for 12 weeks.
  Interventions: Dietary Supplement: Attapulgite
- Placebo (Placebo Comparator): Maltodextrin capsules (0.4-0.5 g) were administered at a dose of 3 capsules twice daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Attapulgite — Participants were administered daily attapulgite (2.5 g) for a duration of 12 weeks.
  Arms: Attapulgite
Dietary Supplement: Placebo — Participants were administered daily maltodextrin (2.5 g) for a duration of 12 weeks.
  Arms: Placebo

SUMMARY:
To explore the safety and efficacy of attapulgite in the treatment of obese individuals or overweight/obese individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Obese individuals:

* Aged 18-60 years, regardless of sex/gender
* BMI≥28.0kg/m2

Overweight or obese individuals with type 2 diabetes:

* Aged 18-60 years, regardless of sex/gender
* BMI≥24.0kg/m2
* HbA1c ≥7.0% and ≤10.0% or the fasting blood glucose ≥7.0 mmol/l and ≤ 13.3 mmol/l at screening
* Stable diabetes treatment for at least 6 months or more

Exclusion Criteria:

* Type 1 diabetes, monogenic diabetes, or diabetes due to pancreatic injury or other secondary diabetes
* Severe diabetic complications within three months before the study initiation, including severe hypoglycemia, diabetic ketoacidosis, or infections
* Use of weight-affecting products within the past three months or planned use during the study
* Weight fluctuation >5 kg or >10% within the past three months
* Obesity or overweight due to endocrine disorders (such as thyroid dysfunction or Cushing's syndrome)
* Uncontrolled hypertension, severe cardiac/hepatic/renal dysfunction
* History of gastrointestinal surgery (such as cholecystectomy) within the past year or non-gastrointestinal surgery within six months, or prior bariatric surgery
* Chronic gastrointestinal disorders (such as recurrent constipation, celiac disease, or food intolerances) or any condition impairing digestion/absorption function
* History of malignant tumors within five years, regardless of whether there is recurrence or metastasis and severe immune dysfunction (such as malignant tumors, HIV/AIDS, immunodeficiency diseases)
* Use of probiotics, prebiotics, or antibiotics within three months prior to enrollment, or alcohol abuse; Consumption of yogurt within two weeks before the study or during the trial period; History of psychiatric or infectious diseases
* Pregnancy, lactation, or plans for pregnancy during the study
* Participation in other clinical trials within the past three months
* Any condition that in the judgement of the investigator precludes participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | "Baseline" "6 weeks" and "12 weeks"
  BMI used to assess body weight relative to height, the unit of BMI is kg/m² (kilograms per square meter).

SECONDARY OUTCOMES:
Weight | "Baseline" "6 weeks" and "12 weeks"
Waist circumference | "Baseline" "6 weeks" and "12 weeks"
Hip circumference | "Baseline" "6 weeks" and "12 weeks"
Waist-to-hip ratio | "Baseline" "6 weeks" and "12 weeks"
Human body fat percentage | "Baseline" and "12 weeks"
  It measured via Lunar iDXA equipment
Human basal metabolic rate | "Baseline" and "12 weeks"
  It measured via Lunar iDXA equipment, including basal metabolic rate, body fat percentage, visceral fat area, subcutaneous fat area, etc.)
Visceral fat mass | "Baseline" and "12 weeks"
  It measured via iDXA equipment
Subcutaneous fat area | "Baseline" and "12 weeks"
  It measured via iDXA equipment
Serum triglycerides | "Baseline" "6 weeks" and "12 weeks"
Serum total cholesterol | "Baseline" "6 weeks" and "12 weeks"
Serum LDL-c | "Baseline" "6 weeks" and "12 weeks"
Serum HDL-c | "Baseline" "6 weeks" and "12 weeks"
Gut microbiome | "Baseline" and "12 weeks"
  including fecal intestinal flora metagenome
Gut metabolites | "Baseline" and "12 weeks"
  In aid of LC/MS and GC/MS technique, etc, we will measure the metabolomics molecular profile in fecal samples before and after treatment.The metabolomics measurement will help to detect the profile of all kinds of lipids species and amino acid species, etc.
Serum metabolites | "Baseline" and "12 weeks"
  In aid of LC/MS and GC/MS technique, etc, we will measure the metabolomics molecular profile in blood samples before and after treatment.The metabolomics measurement will help to detect the profile of all kinds of lipids species and amino acid species, etc.
Fasting serum C peptide levels | "Baseline" "6 weeks" and "12 weeks"
Fasting serum insulin levels | "Baseline" "6 weeks" and "12 weeks"
Fasting blood glucose | "Baseline" "6 weeks" "12 weeks"
  It applies to individuals with overweight or obese type 2 diabetes
Glycated albumin | "Baseline" "6 weeks" and "12 weeks"
  It applies to individuals with overweight or obese type 2 diabetes
Glycated haemoglobin (HbA1c) | "Baseline" "6 weeks" and "12 weeks"
  It applies to individuals with overweight or obese type 2 diabetes
2-hour serum C peptide levels | "Baseline" and "12 weeks"
2-hour serum insulin levels | "Baseline" and "12 weeks"
2-hour blood glucose levels | "Baseline" and "12 weeks"
HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) | "Baseline" "6 weeks" and "12 weeks"
Inflammation markers | "Baseline" "6 weeks" and "12 weeks"
  CRP, IgG, IgA, IgM, IgE
Hepatic function | "Baseline" "6 weeks" and "12 weeks"
  including alanine aminotransferase and aspartate aminotransferase
Serum urea nitrogen | "Baseline" "6 weeks" and "12 weeks"
Serum creatinine | "Baseline" "6 weeks" and "12 weeks"
Serum urinary acid | "Baseline" "6 weeks" and "12 weeks"
Adverse events | 12 weeks
  Safety outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China